CLINICAL TRIAL: NCT03748199
Title: Phase-Ib/IIa Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Orally Inhaled Multiple Doses of POL6014 in Patients With Cystic Fibrosis
Brief Title: Clinical Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of POL6014 in Patients With CF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SNT-I-018
Record Dates: First submitted 2018-11-05; First posted 2018-11-20 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-03

CONDITIONS: Cystic Fibrosis
Keywords: CF; cystic fibrosis; POL6014; neutrophil elastase inhibitor; anti-inflammatory
MeSH Terms: conditions — Cystic Fibrosis | interventions — lonodelestat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POL6014 (Experimental): multiple ascending doses: 80, 160 and 40 mg once or twice daily
  Interventions: Drug: POL6014
- Placebo (Placebo Comparator): Placebo will be administered orally at a dose and frequency matched to POL6014
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: POL6014 — DL1 80 mg cohorts 1A and 1B (80 mg QD and 40 mg BID) DL2 160 mg cohorts 2A and 2B (160 mg QD and 80 mg BID) DL3 40 mg QD cohort C
  DL = dose Level QD= quaque die (once daily) BID= bis in die (twice daily)
  Arms: POL6014
Drug: Placebo — Placebo will be administered orally at a dose and frequency matched to POL6014
  Arms: Placebo

SUMMARY:
"This is a randomised, double-blind, placebo-controlled multi-centre study to investigate safety and tolerability and to provide pharmacokinetic and pharmacodynamics information of orally inhaled multiple doses (80 mg, 160 mg or 320 mg) of the nebulised neutrophil elastase inhibitor POL6014 in patients with Cystic Fibrosis. The controlled inhalation will occur via the eFlow® nebuliser system (manufacturer: PARI Pharma GmbH, Germany)".

ELIGIBILITY:
Inclusion Criteria:

1. Patient has given written informed consent to participation in the trial prior to their enrolment and any trial-related procedure.
2. Male patients or female patients of non-childbearing potential, aged 18 to 55 years, inclusive. Women of non-childbearing potential are defined as those who have no uterus, or ligation of the fallopian tubes, or permanent cessation of ovarian function due to ovarian failure or surgical removal of the ovaries. Documentation of surgical procedure is required for patients who have had a hysterectomy or tubal ligation.
3. Men must agree to practice contraception from start of study medication up to 90 days after the last dose of the study medication.
4. Patient with a diagnosis of CF documented by a compatible clinical or radiographic presentation and laboratory criteria, more specifically, sweat or genetic testing (i.e., presence of the most common genetic defect ΔF 508 or any other mutation that can produce CF).
5. Patient should confirm to produce frequently spontaneous sputum with a frequency of over 3 expectorates per day. Patient should be capable of producing a spontaneous sputum sample at screening (within a time range of approx. 3h during the screening visit).
6. Except for CF and CF-related diseases, no other significant disease as assessed by a screening examination including medical history, physical examination, vital signs, ECG assessment, pulmonary function testing (PFT), and clinical laboratory results. Deviations of clinical laboratory results can be accepted if they are in accordance with the diagnosis of CF and CF-related diseases, supposed they do not indicate a clinical state that is expected to constitute a significant additional risk.
7. Patient must have an FEV1 ≥ 40% of predicted value at screening.
8. Body mass index (BMI) between 16.5 and 30 (both inclusive).
9. Non-smoker or ex-smoker who has stopped smoking for at least one (1) year prior to the Screening Visit.
10. Patient should be willing to refrain from caffeine- or theophylline-containing products within 24 h prior to a clinic visit for a full PK profile.
11. Ability to inhale in an appropriate manner (Patients will be trained to inhale from the eFlow® nebuliser device with a commercially available saline solution at the Screening Visit once informed consent has been obtained).
12. For patients with routine courses of inhaled antibiotics, patients should agree to start routine course of inhaled antibiotic cycle on the same day or not earlier than 3 days before IMP administration.

Exclusion Criteria:

1. Patient with unstable lung disease, as defined by a change in treatment regimen during the preceding two (2) weeks, or a significant new finding on chest radiography (such as, but not limited to, pneumothorax, lobar/segmental collapse or consolidation), or in the opinion of the investigator, patient with a decline in pulmonary status within the last 12 months not considered a part of the usual, chronic progression of CF lung disease. Routine cyclic antibiotic treatment regimens including "off/on" cycles are not considered to be changes to treatment regimens.
2. Patient has had an exacerbation of respiratory symptoms within the past four (4) weeks before screening/randomization that required initiation of a new or altered respiratory therapy, and, in the opinion of the investigator, the patient has not returned to a stable level of health
3. Patient with a history of lung transplantation.
4. Patient with a history of clinically significant renal, hepatic, gastrointestinal,cardiovascular and particularly respiratory disease (excluding CF and CF-related disease).
5. Patient with active gastrointestinal ulcer, history of intracranial bleedings, injuries and other bleedings.
6. Patient, as per assessment of the investigator, with severe hepatic impairment (e.g. laboratory values (ALT, AST > 3 x ULN and total bilirubin > 1.5 x ULN) or Child-Pugh-Class C could be indicative of such condition).
7. ECG abnormalities of clinical relevance (e.g., QTc according to Bazett's formula ≥440 ms, PR >200 ms, or QRS ≥120 ms).
8. Patient with a resting heart rate in supine position <50 bpm, systolic blood pressure <100 mmHg or >140 mmHg, diastolic blood pressure <60 mmHg or >90 mmHg.
9. Proneness to orthostatic dysregulation, fainting, or blackouts.
10. Diagnosis of a tricuspid insufficiency in combination with a mean pulmonary arterial pressure (mPAP) > 25 mmHg, measured by Doppler echography, or, if no tricuspid insufficiency is detectable, any echocardiographic or clinical signs of severe pulmonary heart disease (cor pulmonale) or depending congestive heart failure.
11. History or presence of any malignancy.
12. Positive results in any of the following virology tests: human immunodeficiency virus (HIV) antibodies and antigen, Anti-hepatitis B-core antibody, hepatitis B surface antigen (HbsAg) and anti-hepatitis C virus antibody.
13. Known local or systemic hypersensitivity to any aerosol, medication or food that led to admission to an emergency room.
14. Participation in another clinical study with any investigational medicinal product (IMP) or device, before randomisation, within an interval of 5 half-lives (minimum 4 weeks) from the last use of that investigational drug.
15. Blood or plasma donation of more than 500 mL during the previous month before randomisation, as declared by the patient.
16. Mental condition rendering the patient incapable to understand the nature, scope, and possible consequences of the study.
17. Not willing to comply with all clinical study procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Safety measured by proportion of patients who experience potential clinically significant changes in physical examinations | Baseline through end of treatment (up to 15 days for cohorts 1A/2A/2B, up to 28 days for cohort C)
Safety measured by number of patients with changes in laboratory assessments (clinical chemistry, haematology, urinanalysis) | Baseline through end of treatment (up to 15 days for cohorts 1A/2A/2B, up to 28 days for cohort C)
Safety measured by number of patients with changes in vital signs (blood pressure, pulse, respiratory rate and body temperature) | Baseline and pre-dose through end of treatment (up to 15 days for cohorts 1A/2A/2B, up to 28 days for cohort C)
Safety measured by number of patients with changes in ECG parameters (heart rythm, ventricular rate, PR interval, QRS duration, Qt and QTc) | Baseline and pre-dose through end of treatment (up to 15 days for cohorts 1A/2A/2B, up to 28 days for cohort C)
Safety measured by occurrence and severity of adverse events | Baseline through end of treatment (up to 15 days for cohorts 1A/2A/2B, up to 28 days for cohort C)
Safety measured by proportion of subjects who experience local irritation of the nose or pharynx by visual inspection | Baseline through end of treatment (up to 15 days for cohorts 1A/2A/2B, up to 28 days for cohort C)
Safety measured by proportion of patients who experience bronchospasm | Baseline through end of treatment (up to 15 days for cohorts 1A/2A/2B, up to 28 days for cohort C)
Safety measured by changes in lung function parameters (FEV1, FVC) | Baseline and pre-dose through end of treatment (up to 15 days for cohorts 1A/2A/2B, up to 28 days for cohort C)
Safety measured by changes in oxygen saturation in peripheral blood as measured by pulse oximetry | Baseline through end of treatment (up to 15 days for cohorts 1A/2A/2B, up to 28 days for cohort C)
Tolerability assessed by the number of patients who discontinue the study treatment prematurely due to Adverse Events | Baseline through end of treatment (up to 15 days for cohorts 1A/2A/2B, up to 28 days for cohort C)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) for POL6014 and metabolites in plasma, sputum and urine | At defined timepoints (Day1, Day 2, Day 8, Day 14, Day 15, Day 16)
  Concentration of POL6014 and relevant metabolites measured in plasma, sputum and urine

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Charité - Uniklinik Berlin, Klinik für Pädiatrie,Pneumologie, Immunologie, Erwachsenene-Mucoviszidose, Berlin
  - Ruhrlandklinik Westdeutsches Lungenzentrum, Essen
  - IKF Pneumologie GmbH & Co. KG, Institut für klinische Forschung Pneumologie, Frankfurt
  - Inamed GmbH, clinical unit, Gauting